CLINICAL TRIAL: NCT00206518
Title: A Randomized Multicenter Trial of Neoadjuvant Taxotere (T) and Adriamycin/Cytoxan (Ac): A Validation
Brief Title: Taxotere and Adriamycin/Cytoxan (AC) Validation in Breast Cancer Patients
Acronym: TACAC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mothaffar Rimawi (Other)
Collaborators: Baylor College of Medicine (Other)
Responsible Party: Sponsor-Investigator, Mothaffar Rimawi, Medical Director, Baylor Breast Care Center
Organization: Baylor Breast Care Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H 16039
Record Dates: First submitted 2005-09-14; First posted 2005-09-21 (Estimated); Results first posted 2017-06-06 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Breast Cancer
Keywords: Breast; Cancer; Taxotere; AC; Validation; Neoadjuvant
MeSH Terms: conditions — Breast Neoplasms; Neoplasms | interventions — Docetaxel; Doxorubicin; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A: Taxotere/Docetaxel (Experimental): Chemotherapy In Arm A, patients will receive single agent Taxotere (100 mg/m2) every 3 weeks for 4 cycles before surgery. Primary surgery will then be conducted, if operable, following completion of neoadjuvant treatment. This will be followed by standard adjuvant AC (doxorubicin 60 mg/m2 and cyclophosphamide 600 mg/m2, every 3 weeks) for 4 cycles. For patients whose BSA is greater than 2.0 m2, the Adriamycin dosage will be calculated using BSA = 2.0 m2. This is done in order to minimize Adriamycin-induced cardiotoxicity.
  Interventions: Drug: Taxotere/Docetaxel; Drug: doxorubicin
- B: AC Adriamycin/Cytoxan (Experimental): In Arm B, patients will receive AC (doxorubicin 60 mg/m2 and cyclophosphamide 600 mg/m2, every 3 weeks) for 4 cycles before surgery. For patients whose BSA is greater than 2.0 m2, the Adriamycin dosage will be calculated using BSA = 2.0 m2. Primary surgery will then be conducted, if operable, following completion of neoadjuvant treatment. This will be followed by 4 cycles of single agent Taxotere (100 mg/m2) every 3 weeks.
  Interventions: Drug: Adriamycin/Cytoxan

INTERVENTIONS:
Drug: Taxotere/Docetaxel — Taxotere
  Other Names: docetaxel
  Arms: A: Taxotere/Docetaxel
Drug: Adriamycin/Cytoxan — Adriamycin/Cytoxan
  Other Names: doxorubicin
  Arms: B: AC Adriamycin/Cytoxan
Drug: doxorubicin — AC (doxorubicin 60 mg/m2 and cyclophosphamide 600 mg/m2, every 3 weeks) for 4 cycles before surgery.
  Other Names: AC, ADRIAMYCIN/CYTOXAN
  Arms: A: Taxotere/Docetaxel

SUMMARY:
The purpose of this study is to learn if the biomarker information obtained (learned or received) from the earlier studies can tell us whether or not Taxotere and/or Adriamycin/Cytoxan can cause tumors to become smaller.

DETAILED DESCRIPTION:
Large clinical trials have confirmed the value of systemic adjuvant therapy in decreasing the risk of recurrence and death in patients with early breast cancer. However, the need to identify breast cancer patients who will benefit from adjuvant therapy, while sparing others from the side effects of futile treatment, is spurring research into predictive markers of chemotherapy sensitivity and resistance. In the adjuvant setting, extremely large trials and long follow-up would be required to prospectively validate the predictive value of biomarkers of chemotherapy sensitivity or resistance. In part this is because response is not directly observable. Preoperative chemotherapy for large tumors (>3cm) or inoperable breast cancer is well established and is the standard of care for locally advanced breast cancer. Data from large series of patients have demonstrated that preoperative (neoadjuvant) chemotherapy leads to significant reduction of tumor size (downstaging) and improves both the rate and the cosmetic results of breast- conserving surgery. The degree of response to neoadjuvant therapy has been shown to predict improved overall survival. This is therefore an attractive setting to study predictors of response because tissue is accessible from pre- therapeutic biopsies and tumor response is directly observable.

In an early proof-of-principle pilot study of single agent neoadjuvant docetaxol, we identified a predictive gene expression pattern, and, using leave-one-cross validation, a method of internal validation, we demonstrated that the pattern was likely to accurately discriminate between responders and non-responders (Chang, J.C., et al., Gene expression profiling for the prediction of therapeutic response to docetaxel in patients with breast cancer. Lancet, 2003. 362(9381): p. 362-9). A similar pilot study of neoadjuvant AC undertaken by a collaborator in the UK suggests that different profiles will be predictive for AC response.

In order to definitively determine predictive patterns for both regimens (T and AC) using improved technology for RNA preparation and a larger, more comprehensive gene expression array, we undertook a randomized Phase II trial of these two widely used regimens (Protocol H-11624 - A RANDOMIZED MULTICENTER TRIAL OF NEOADJUVANT TAXOTERE AND ADRIAMYCIN/CYTOXAN (AC): A BIOLOGIC CORRELATIVE STUDY). The trial is nearing completion, having recruited more than 90 patients out of an expected 120 patients. To date, the risks associated with this study have been modest, and there have been no unexpected adverse events. The laboratory work is well underway and gives every indication that clinically useful classifiers to predict treatment efficacy will result.

ELIGIBILITY:
Inclusion Criteria:

1. All patients must be female.
2. Signed informed consent.
3. Primary breast cancers must be of clinical and/or radiologic size >3 cm, and deemed surgically operable.
4. Negative serum pregnancy test (bHCG) within 7 days of starting study, if of child-bearing potential.
5. Adequate bone marrow function:

   * Hematocrit of greater than 30%,
   * total neutrophil count must be >1.5 x 10^9/L and
   * platelets of > 100 x 10^9/L prior to the start of any cycle.
6. Renal function tests:

   * creatinine within 1.5 times of the institution's upper limit of normal (ULN).
7. Liver function tests:

   * Total serum bilirubin within ULN, and
   * liver transaminases within 2.5 times ULN, and
   * alkaline phosphatase within 5 times ULN.
8. Electrocardiogram showing no acute ischemic changes.
9. Performance status (World Health Organization [WHO] scale) <2.
10. Age > 18 years.
11. Patients older than 70 years of age should have left ventricular ejection fraction within ULN by multigated acquisition scan (MUGA) or 2D echocardiogram.

Exclusion Criteria:

1. Patients with metastatic breast cancer.
2. Pregnancy or unwillingness to use a reliable contraceptive method in women of child-bearing potential.
3. Women who are lactating or breastfeeding.
4. Severe underlying chronic illness or disease.
5. Peripheral neuropathy - grade 2 or greater.
6. Patients on other investigational drugs while on study will be excluded.
7. Severe or uncontrolled hypertension, history of congestive heart failure, acute myocardial infarction, or severe coronary arterial disease.
8. Prior taxane or anthracycline chemotherapy for malignancy.
9. Patients with a history of severe hypersensitivity reaction to Taxotere or other drugs formulated with polysorbate 80.
10. No previous or current malignancies at other sites within the last 5 years, with exception of adequately treated cone-biopsied in situ carcinoma of the cervix uteri and basal or squamous cell carcinoma of the skin.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2004-09; Primary Completion 2016-10 (Actual); Study Completion 2016-10-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mothaffar Rimawi, MD, Principal Investigator — Baylor Breast Center
Locations (1):
- Baylor Breast Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | A: Taxotere/Docetaxel | B: AC Adriamycin/Cytoxan
Started | 83 | 84
Completed | 73 | 78
Not Completed | 10 | 6
Not completed — Lack of Efficacy | 6 | 4
Not completed — Adverse Event | 2 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Protocol Violation | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A: Taxotere/Docetaxel | B: AC Adriamycin/Cytoxan | Total
Number analyzed (Participants) | 83 | 84 | 167
Age, Customized [Number; unit: participants]
  <=50 years | 56 | 49 | 105
  >50 years | 27 | 35 | 62
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 84 | 167
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 21 | 27 | 48
  Hispanic | 35 | 34 | 69
  Black | 24 | 18 | 42
  Asian | 3 | 5 | 8

OUTCOME MEASURES:

1. Primary Outcome: Pathological Tumor Response to Neoadjuvant Chemotherapy (Taxotere and AC)
Description: The patients' pathological response were assessed using Chevalier's system which graded the responses into Chevalier 1, 2, 3A, 3B, 3C, 3D, and 4, defined as:
  1. Disappearance of all tumor either on macroscopic or microscopic assessment in both the breast and LN (pCR)
  2. Presence of in situ carcinoma in the breast. No invasive tumor in breast and no tumor in LN (pCR)
  3. Presence of invasive cancer with stromal alteration such as sclerosis or fibrosis (pPR) 3A: Subjectively > 75% therapeutic effect 3B: Subjectively between 50% - 75% therapeutic effect 3C: Subjectively between 25% - 50% therapeutic effect 3D: Subjectively < 25% therapeutic effect OR Grade 4
  4. No or few modification of tumoral appearance (pNR).
Time Frame: 10 years
Measure: Number; unit: participants
Arm/Group | A: Taxotere/Docetaxel | B: AC Adriamycin/Cytoxan
Number analyzed (Participants) | 83 | 84
participants
  1 | 3 | 9
  2 | 2 | 1
  3A | 18 | 15
  3B | 15 | 18
  3C | 18 | 15
  3D | 10 | 8
  4 | 3 | 0
  N/A | 14 | 18

2. Secondary Outcome: Disease Relapse
Description: Data associated with relapse and progression will be obtained over the course of 10 years. Relapse/progression was defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 10 years
Measure: Number; unit: participants
Arm/Group | A: Taxotere/Docetaxel | B: AC Adriamycin/Cytoxan
Number analyzed (Participants) | 83 | 84
participants
  relapsed | 24 | 25
  not relapsed | 59 | 59

3. Secondary Outcome: Overall Survival
Time Frame: 10 years
Measure: Number; unit: participants
Arm/Group | A: Taxotere/Docetaxel | B: AC Adriamycin/Cytoxan
Number analyzed (Participants) | 83 | 84
participants
  deceased | 16 | 19
  alive | 67 | 65

ADVERSE EVENTS:
Arm/Group | A: Taxotere/Docetaxel | B: AC Adriamycin/Cytoxan
Serious Adverse Events (participants affected / at risk) | 12/83 | 5/84
Other Adverse Events (participants affected / at risk) | 13/83 | 3/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A: Taxotere/Docetaxel (N=83) | B: AC Adriamycin/Cytoxan (N=84)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 1 (1)
ALLERGIC/REACTION (Immune system disorders) | 1 (1) | 0 (0)
NEUTROPENIA (Blood and lymphatic system disorders) | 8 (12) | 3 (6)
FEVER (General disorders) | 2 (2) | 1 (1)
GASTRITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
INFECTION (Infections and infestations) | 4 (6) | 1 (1)
RENAL FAILURE (Renal and urinary disorders) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A: Taxotere/Docetaxel (N=83) | B: AC Adriamycin/Cytoxan (N=84)
NEUTROPENIA (Blood and lymphatic system disorders) | 13 (20) | 3 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes